CLINICAL TRIAL: NCT01683006
Title: Influence of Skeletal Muscle Paralysis on Metabolism in Hypothermic Patients After Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ulrike Holzinger, MD, Assoc Prof, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 753/2009UH
Record Dates: First submitted 2012-04-08; First posted 2012-09-11 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Critical Illness; Cardiac Arrest
MeSH Terms: conditions — Critical Illness; Heart Arrest | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuromuscular blocker group (Active Comparator): Continuous application of neuromuscular blockers during therapeutic hypothermia.
  Bolus application of placebo in case of shivering.
  Interventions: Drug: Rocuronium
- Placebo group (Placebo Comparator): Continuous application of placebo during therapeutic hypothermia.
  Bolus application of neuromuscular blockers in case of shivering.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rocuronium — Continuous application of Rocuronium (0.5 mg/kg body weight/hour).
  Bolus application of placebo in case of shivering.
  Arms: Neuromuscular blocker group
Drug: Placebo — Continuous application of placebo during therapeutic hypothermia.
  Bolus application of Rocuronium (0.5 mg/kg body weight) in case of shivering.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate the impact of muscle relaxing drugs on the energy rate during hypothermia after cardiac arrest.

DETAILED DESCRIPTION:
Mild hypothermia improves neurological outcome after cardiac arrest. Neuromuscular blockers are in use, together with analgesia and sedation, during the cooling process in many centers to prevent shivering. However, neuromuscular blockers are accused to be associated with various side effects causing serious harm and/or leading to prolonged ICU stay. Furthermore, the use of neuromuscular blockers may mask epileptic activity. Therefore, the advantages and disadvantages of neuromuscular blockers during therapeutic hypothermia need to be re-evaluated.

Aim of this study is to investigate if continuous application of neuromuscular blockers is necessary to prevent shivering and thereby avoiding an increase in energy expenditure in patients during therapeutic hypothermia and rewarming after cardiac arrest (initial 72h).

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving mild therapeutic hypothermia after cardiac arrest of presumed cardiopulmonary origin

Exclusion Criteria:

* age < 18
* cardiac arrest >6 hours before admittance at the hospital
* patients with known or clinically apparent pregnancy
* patients who reach our hospital with a body temperature below 35°C
* patients with known allergic reactions against rocuronium
* patients with a history of myasthenia gravis
* patients with obvious intoxication
* wards of the state/prisoners
* patients with known epileptic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change of resting energy expenditure compared to baseline at 33C° | initial 72h after cardiac arrest at defined temperatures or timepoints: 1) 33°C 2) 34.5°C 3) 36 °C 4) 36.5 - 37.5 °C 5) after 48-72h
  resting energy expenditure will be assessed with indirect calorimetry at different measurement time points:
  1. 12-24 h after initiation of mild hypothermia (33C°)
  2. during warming up (at 34.5°C)
  3. during warming up (at 36°C)
  4. during warming up (at 36.5°C - 37.5°C)
  5. normal Temperature, after 48 - 72 h after initiation of mild hypothermia

SECONDARY OUTCOMES:
Change of substrate oxidation rate (protein, fat and glucose) compared to baseline at 33C° | initial 72h after cardiac arrest at defined temperatures or timepoints: 1) 33°C 2) 34.5°C 3) 36 °C 4) 36.5 - 37.5 °C 5) after 48-72h
  substrate oxidation rates will be assessed with indirect calorimetry at different measurement time points:
  1. 12-24 h after initiation of mild hypothermia (33C°)
  2. during warming up (at 34.5°C)
  3. during warming up (at 36°C)
  4. during warming up (at 36.5°C - 37.5°C)
  5. at normal Temperature, after 48 - 72 h after initiation of mild hypothermia

OTHER OUTCOMES:
Difference in resting energy expenditure between patients with favorable and unfavorable outcome | initial 72h after cardiac arrest at defined temperatures or timepoints: 1) 33°C 2) 34.5°C 3) 36 °C 4) 36.5 - 37.5 °C 5) after 48-72h
  resting energy expenditure will be assessed with indirect calorimetry at different measurement time points:
  1. 12-24 h after initiation of mild hypothermia (33C°)
  2. during warming up (at 34.5°C)
  3. during warming up (at 36°C)
  4. during warming up (at 36.5°C - 37.5°C)
  5. normal Temperature, after 48 - 72 h after initiation of mild hypothermia
Difference in substrate metabolism between patients with favorable and unfavorable outcome | initial 72h after cardiac arrest at defined temperatures or timepoints: 1) 33°C 2) 34.5°C 3) 36 °C 4) 36.5 - 37.5 °C 5) after 48-72h
  substrate oxidation rates will be assessed with indirect calorimetry at different measurement time points:
  1. 12-24 h after initiation of mild hypothermia (33C°)
  2. during warming up (at 34.5°C)
  3. during warming up (at 36°C)
  4. during warming up (at 36.5°C - 37.5°C)
  5. at normal Temperature, after 48 - 72 h after initiation of mild hypothermia

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Holzinger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University Vienna, Vienna, Austria